CLINICAL TRIAL: NCT01778257
Title: Mate Extract Supplementation Reduces Body and Abdominal Fat in Obese Korean Subjects
Brief Title: Efficacy and Safety of Mate Extracts on Decrement of Body and Abdominal Fat in Obese Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chonbuk National University Hospital (Other)
Collaborators: GS Engineering & Construction (Unknown)
Responsible Party: Principal Investigator, Min-Gul Kim, MD, Clinical Assistant Professor, Chonbuk National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CUH_2011_GS_MATE
Record Dates: First submitted 2012-12-07; First posted 2013-01-29 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Obesity
Keywords: Mate extracts; Obesity; abdominal fat
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mate extracts group (Experimental): Mate extract(3150 mg/day)for 12 weeks
  Interventions: Dietary Supplement: Mate extract
- Placebo group (Placebo Comparator): Placebo (3150 mg/day) for 12 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Mate extract — Mate is a South American herb that is traditionally prepared as a tea and used, among others, for weight reduction.
  Other Names: Extracts of Ilex paraguariensis A. St.-Hil.
  Arms: Mate extracts group
Dietary Supplement: Placebo — Amount and calorie of placebo are same with Mate extracts.
  Arms: Placebo group

SUMMARY:
Obesity is a major health issue worldwide; there is a constant raise in obesity related death each year.

DETAILED DESCRIPTION:
The primary aim of the study was to investigate the effect of Mate extracts in Korean subjects on body fat and abdominal fat, double blind, placebo-controlled clinical trial.

Thirty obesity subjects with BMI ≥ 25 kg/㎡ and waist-hip ratio (WHR)≥ 0.90 for men and ≥ 0.85 for women were for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers aged 19 to 65 years
* 25 kg/m2 ≤ BMI ≥35 kg/m2
* Ability to give informed consent

Exclusion Criteria:

* Significant variation in weight (more 10%) in the past 3 month
* Cardiovascular disease, neurologic or psychiatric disease, renal, pulmonary and hepatic abnormalities
* History of disease that could interfere with the test products or impede their absorption, such as gastrointestinal disease (Crohn's disease) or gastrointestinal surgery (a caesum or enterocele surgery are included)
* Laboratory test, medical or psychological conditions deemed by the investigators to interfere with successful participation in the sutdy
* Allergic or hypersensitive to any of the ingredients in the test products
* Pregnancy or breast feeding
* Used antipsychosis drugs therapy within past 2 months
* History of alcohol or substance abuse (21 units/week over)
* Participation in any other clinical trials within past 3 months

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-10; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Changes in body and abdominal fat | body fat: baseline, 6 weeks and 12 weeks, abdominal fat of CT: baseline and 12 weeks

SECONDARY OUTCOMES:
Changes in anthropometric parameters(weight, BMI, waist and hip circumference) | baseline, 6 weeks and 12 weeks
Changes in blood lipid profile(total cholesterol, triglyceride, HDL-cholesterol, LDL-cholesterol, free fatty acid) | baseline, 6 weeks and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Min-Gul Kim, MD, Principal Investigator — Chonbuk National University Hospital

REFERENCES:
- [Derived] Kim SY, Oh MR, Kim MG, Chae HJ, Chae SW. Anti-obesity effects of Yerba Mate (Ilex Paraguariensis): a randomized, double-blind, placebo-controlled clinical trial. BMC Complement Altern Med. 2015 Sep 25;15:338. doi: 10.1186/s12906-015-0859-1. PMID 26408319